CLINICAL TRIAL: NCT04948086
Title: Blood Pressure Lowering Effect of B-vitamins in Adults With a Genetic Pre-disposition to Elevated Blood Pressure.
Brief Title: Blood Pressure and Central Haemodynamics in Healthy Adults Stratified by MTHFR Genotype
Acronym: RAFA Obs
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Other Study IDs: REC/11/0081 Obs
Record Dates: First submitted 2021-06-11; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; MTHFR; Methylenetetrahydrofolate Reductase; Central Hemodynamics; Riboflavin; Folic Acid; Folate Polymorphism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, washed red cells, whole blood, whole blood in ascorbic acid (1 in 10 dilution), buffy coat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TT MTHFR genotype
- Non-TT (i.e. CC/CT) MTHFR genotype

SUMMARY:
Approximately 12% of the world's population have a have a common C677T polymorphism in the gene encoding the folate metabolising enzyme, methylenetetrahydrofolate reductase (MTHFR). Homozygosity for the polymorphism (TT genotype) appears to result in an increased requirement for the B-vitamins folic acid and riboflavin and more importantly results in an increased risk of developing high blood pressure (BP). Previous work from our Centre has demonstrated significantly higher BP in those with the TT genotype. This work has been conducted in cohorts with premature cardiovascular disease (CVD) and hypertension without overt CVD, but the effect in younger, healthier individuals is unexplored. To date our studies have also focused on BP as the primary outcome, but newer markers of vascular health including central pressure and hemodynamics have emerged as superior prognostic indicators of CVD. The effect of the TT genotype on these measures is thus an important area for investigation and may help us understand the mechanism linking the genotype with BP, which is currently unknown. As adults with the TT genotype appear to have increased requirements for riboflavin and folic acid, and BP in TT adults appears to be riboflavin dependent, the influence of these vitamins on central measures is an area for consideration. Study Design This is an observational study investigating the blood pressure profiles of healthy adults aged 18-65 years, stratified by MTHFR genotype. Apparently healthy adults will be recruited from workplaces and the general community across Northern Ireland and screened for the polymorphism via buccal swab. Those with the TT genotype and a similar number of non-TT (i.e. CC/CT) genotype individuals will be contacted and asked to come to attend a one-off appointment. Brachial BP will be assessed by an electronic BP monitor, central BP and central haemodynamics (augmentation index, augmentation pressure and pulse wave velocity) will be assessed by SphygmoCor XCEL. In addition, anthropometric measurements, health and lifestyle information and a blood sample will be obtained. Data will be statistically analysed using SPSS software to if determine differences between gentoype groups exist.

ELIGIBILITY:
Inclusion Criteria:

* Pre-screened for MTHFR 677TT genotype
* Aged at least 18 years old

Exclusion Criteria:

* Younger than 18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Blood pressure | One day, one measurement
  Office blood pressure

SECONDARY OUTCOMES:
Brachial blood pressure | One day, one measurement
  Measured using SphygmoCor device
Central blood pressure | One day, one measurement
  Measured using SphygmoCor device
Pulse wave analysis | One day, one measurement
  Measured using SphygmoCor device
Pulse wave velocity | One day, one measurement
  Measured using SphygmoCor device
Riboflavin status | One day, one measurement
  Measured by by EGRac
Folate status | One day, one measurement
  Measured by microbiological assay
PLP status | One day, one measurement
  Measured by HPLC
Homocysteine status | One day, one measurement
  Measured by GCMS
One-carbon metabolite status | One day, one measurement
  Measured by GCMS-MS

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom